CLINICAL TRIAL: NCT07341854
Title: Effect of Intravenous Dexamethasone Palmitate on Postoperative Pain Prevention
Brief Title: Dexamethasone Palmitate for Postoperative Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Beijing Ditan Hospital (Other); Beijing Electric Power Hospital (Other)
Responsible Party: Principal Investigator, Fang Luo, Director of Department of Pain Management, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KY2025-041-02-04
Record Dates: First submitted 2025-12-14; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Pain, Postoperative; Dexamethasone Palmitate
MeSH Terms: conditions — Pain, Postoperative | interventions — dexamethasone 21-palmitate; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexamethasone palmitate group (Experimental): Patients assigned to the dexamethasone palmitate group will receive an intravenous injection of 8 mg dexamethasone palmitate after induction of anaesthesia but prior to surgical incision.
  Interventions: Drug: dexamethasone palmitate
- Dexamethasone group (Active Comparator): Patients in the dexamethasone group will receive an intravenous injection of 8 mg dexamethasone after induction of anaesthesia but prior to surgical incision.
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: dexamethasone palmitate — Patients assigned to the dexamethasone palmitate group will receive an intravenous injection of 8 mg dexamethasone palmitate after induction of anaesthesia but prior to surgical incision.
  Arms: Dexamethasone palmitate group
Drug: Dexamethasone — Patients in the dexamethasone group will receive an intravenous injection of 8 mg dexamethasone after induction of anaesthesia but prior to surgical incision.
  Arms: Dexamethasone group

SUMMARY:
Postoperative pain remains highly prevalent and inadequately managed in a significant proportion of surgical patients, often leading to delayed recovery, increased opioid consumption, and potential progression to chronic pain. While perioperative systemic dexamethasone is used for its anti-inflammatory and opioid-sparing effects, its efficacy is inconsistent, and concerns regarding systemic side effects persist. Dexamethasone palmitate, a novel lipophilic prodrug formulated as nanoparticle emulsion, leverages the enhanced permeability and retention effect to target inflammatory sites selectively, potentially offering superior anti-inflammatory and analgesic efficacy with reduced systemic exposure. This trial aims to evaluate whether preoperative intravenous dexamethasone palmitate is more effective than conventional dexamethasone in preventing moderate-to-severe postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years.
2. Scheduled for a range of surgeries under general anesthesia, including both minimally invasive procedures (such as video-assisted thoracoscopic surgery and laparoscopy) and open surgeries (such as thoracotomy, laparotomy, spinal surgery, total joint replacement, and mastectomy).
3. Capacity to comprehend the study procedures and assessment scales, and communicate effectively with research staff.
4. Willingness to participate voluntarily and provide written informed consent.

Exclusion Criteria:

1. Known hypersensitivity to dexamethasone or its excipients.
2. Systemic glucocorticoid therapy within 3 months prior to enrolment.
3. History of severe cardiovascular disease, hepatic or renal failure, or systemic rheumatic disease (e.g., rheumatoid arthritis, ankylosing spondylitis, systemic lupus erythematosus).
4. Coexisting chronic pain at enrolment.
5. Uncontrolled diabetes mellitus or active systemic infection.
6. Significant cognitive impairment or severe psychiatric disorder.
7. Pregnancy or lactation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 446 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
The percentage of participants experiencing moderate to severe pain | 24 hours after surgery
  The percentage of participants experiencing moderate to severe pain (Visual Analog Scale [VAS]>30 mm)

SECONDARY OUTCOMES:
Cumulative opioid consumption | At 6, 24, 48, and 72 hours postoperatively
  Cumulative opioid consumption, expressed as morphine milligram equivalents (MME)
The total consumption of supplemental oxycodone/paracetamol tablets | At 6, 24, 48, and 72 hours postoperatively
  The total consumption of supplemental oxycodone/paracetamol tablets, expressed as the number of tablets
The proportion of participants experiencing moderate to severe pain | At 6, 24, 48, and 72 hours postoperatively
  The proportion of participants experiencing moderate to severe pain at rest and during passive movement (e.g., coughing, deep breathing, or following a 5 m walk test)
Time to first patient-controlled analgesia (PCA) bolus request | Within the first 72 hours postoperatively
  Time to first PCA bolus request
Participant satisfaction with pain management | At 6, 24, 48, and 72 hours postoperatively and at discharge
  Using a 0-10 point numerical rating scale (NRS) (0 = very dissatisfied to 10 = most satisfied imaginable)
Incidences of postoperative nausea and vomiting (PONV) | At 6, 24, 48, and 72 hours after surgery
  PONV is defined as any nausea, vomiting, retching, or combination thereof. Nausea refers to an unpleasant sensation associated with the urge to vomit; vomiting is defined as the forceful expulsion of gastric contents; and retching indicates an involuntary attempt to vomit without producing gastric contents.
Quality of recovery | At 24, 48, and 72 hours postoperatively, as well as at 1 month after surgery.
  Quality of recovery will be measured using the 15-item quality of recovery scoring system [QoR-15] questionnaire. The total score ranges from 0 to 150, where higher scores indicate a better quality of recovery.
Length of hospital stay | From the date of hospital admission to the date of discharge, assessed throughout the hospitalization period (up to 1 month).
  Length of hospital stay was defined as the number of days from the date of hospital admission to the date of discharge.
Incidence of postoperative adverse events | Within one month after surgery
  This outcome measure assesses the occurrence of specified safety events within one month after surgery. The number of participants experiencing any of the following confirmed events will be recorded and reported based on clinical examination, medical record review, and necessary laboratory tests: hypotension, hypertension, gastrointestinal ulcers, poor wound healing, surgical site infection, urinary retention, and hyperglycemia. Data will be aggregated and reported as event frequency and participant count.

CONTACTS AND LOCATIONS:
Locations (1):
- Fang Luo, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
All personal identifiers will be stored securely by the principal investigator, separate from the pseudonymized study data. Access is restricted to the research team, and all published findings will be based on anonymized data aggregates.

REFERENCES:
- [Background] Gan TJ, Habib AS, Miller TE, White W, Apfelbaum JL. Incidence, patient satisfaction, and perceptions of post-surgical pain: results from a US national survey. Curr Med Res Opin. 2014 Jan;30(1):149-60. doi: 10.1185/03007995.2013.860019. Epub 2013 Nov 15. PMID 24237004
- [Background] Apfelbaum JL, Chen C, Mehta SS, Gan TJ. Postoperative pain experience: results from a national survey suggest postoperative pain continues to be undermanaged. Anesth Analg. 2003 Aug;97(2):534-540. doi: 10.1213/01.ANE.0000068822.10113.9E. PMID 12873949
- [Background] Liu Y, Xiao S, Yang H, Lv X, Hou A, Ma Y, Jiang Y, Duan C, Mi W; CAPOPS Group. Postoperative pain-related outcomes and perioperative pain management in China: a population-based study. Lancet Reg Health West Pac. 2023 Jun 10;39:100822. doi: 10.1016/j.lanwpc.2023.100822. eCollection 2023 Oct. PMID 37927993
- [Background] Gandhi K, Heitz JW, Viscusi ER. Challenges in acute pain management. Anesthesiol Clin. 2011 Jun;29(2):291-309. doi: 10.1016/j.anclin.2011.04.009. PMID 21620344
- [Background] Gan TJ. Poorly controlled postoperative pain: prevalence, consequences, and prevention. J Pain Res. 2017 Sep 25;10:2287-2298. doi: 10.2147/JPR.S144066. eCollection 2017. PMID 29026331
- [Background] Tammachote N, Kanitnate S. Intravenous Dexamethasone Injection Reduces Pain From 12 to 21 Hours After Total Knee Arthroplasty: A Double-Blind, Randomized, Placebo-Controlled Trial. J Arthroplasty. 2020 Feb;35(2):394-400. doi: 10.1016/j.arth.2019.09.002. Epub 2019 Sep 7. PMID 31587982
- [Background] Kitcharanant N, Leurcharusmee P, Atthakomol P, Jingjit W. Perioperative intravenous dexamethasone did not reduce the severity of persistent postsurgical pain after total knee arthroplasty: a prospective, randomized, double-blind, placebo-controlled trial. J Orthop Surg Res. 2024 Dec 19;19(1):854. doi: 10.1186/s13018-024-05362-y. PMID 39702151
- [Background] Lorscheider M, Tsapis N, Ur-Rehman M, Gaudin F, Stolfa I, Abreu S, Mura S, Chaminade P, Espeli M, Fattal E. Dexamethasone palmitate nanoparticles: An efficient treatment for rheumatoid arthritis. J Control Release. 2019 Feb 28;296:179-189. doi: 10.1016/j.jconrel.2019.01.015. Epub 2019 Jan 16. PMID 30659904
- [Background] Hui H, Miao H, Qiu F, Lin Y, Li H, Zhang Y, Jiang B. Adjunctive dexamethasone palmitate use for intercostal nerve block after video-assisted thoracoscopic surgery: A prospective, randomized control trial. Heliyon. 2023 Aug 22;9(9):e19156. doi: 10.1016/j.heliyon.2023.e19156. eCollection 2023 Sep. PMID 37662806